CLINICAL TRIAL: NCT00565188
Title: Application of Adenosine 5'-Triphosphate (ATP) Infusions in Palliative Home Care
Brief Title: Application of ATP Infusions in Palliative Home Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 01-092.3; ZonMW 1135.0010
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2007-11

CONDITIONS: Cancer; Palliative Care; Survival; Quality of Life
MeSH Terms: conditions — Neoplasms | interventions — Adenosine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental)
  Interventions: Drug: Adenosine 5'-triphosphate
- C (No Intervention)

INTERVENTIONS:
Drug: Adenosine 5'-triphosphate — Weekly ATP infusions (in total 8 infusions) during 8 - 12 hours in a maximum dose of 50 mcg/kg.min
  Arms: I

SUMMARY:
Palliative care in cancer aims at alleviating the suffering of patients. A previous study in patients with advanced non-small-cell lung cancer showed that adenosine 5'-triphosphate (ATP) infusions had a favourable effect on fatigue, appetite, body weight, muscle strength, functional status, quality of life, and survival. Based on these promising results, the present study was designed 1. To evaluate whether the beneficial effects of ATP administration observed in patients with advanced lung cancer would also be present in pre-terminal cancer patients of different tumour types, and 2. To test the feasibility of application of ATP infusions in a home care setting.

ELIGIBILITY:
Inclusion Criteria:

* cytologically or histologically confirmed cancer
* medical treatment options restricted to supportive care
* a life expectancy < 6 months
* World Health Organization (WHO) performance status 1 or 2
* suffering from at least one of the following complaints: fatigue, weight loss > 5% over the last 6 months, or anorexia

Exclusion Criteria:

* symptomatic angina pectoris
* symptomatic heart failure
* any form of atrioventricular (AV) block (assessed by electrocardiogram)
* life expectancy < 4 weeks
* concurrent palliative chemotherapy
* cognitive dysfunction, and other diseases hampering adequate follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Survival Physical restriction Fatigue Quality of life | 0-8 weeks

SECONDARY OUTCOMES:
Appetite Nutritional intake Body height Body weight Triceps skin fold thickness Mid-upper arm circumference Strength of elbow flexor and knee extensor muscles Handgrip strength Process evaluation | 0-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: P.C. Dagnelie, PhD, Principal Investigator — Maastricht University - Department of Epidemiology
Locations (5):
- Netherlands (5):
  - Maxima Medical Center, Eindhoven
  - Catharina Hospital Eindhoven, Eindhoven
  - Atrium MC, Heerlen
  - Maastricht University Hospital, Maastricht
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] Agteresch HJ, Dagnelie PC, van der Gaast A, Stijnen T, Wilson JH. Randomized clinical trial of adenosine 5'-triphosphate in patients with advanced non-small-cell lung cancer. J Natl Cancer Inst. 2000 Feb 16;92(4):321-8. doi: 10.1093/jnci/92.4.321. PMID 10675381
- [Background] Agteresch HJ, Rietveld T, Kerkhofs LG, van den Berg JW, Wilson JH, Dagnelie PC. Beneficial effects of adenosine triphosphate on nutritional status in advanced lung cancer patients: a randomized clinical trial. J Clin Oncol. 2002 Jan 15;20(2):371-8. doi: 10.1200/JCO.2002.20.2.371. PMID 11786563
- [Background] Agteresch HJ, Burgers SA, van der Gaast A, Wilson JH, Dagnelie PC. Randomized clinical trial of adenosine 5'-triphosphate on tumor growth and survival in advanced lung cancer patients. Anticancer Drugs. 2003 Sep;14(8):639-44. doi: 10.1097/00001813-200309000-00009. PMID 14501386